CLINICAL TRIAL: NCT06219668
Title: The Effect of Omentopexy and Clips on the Staple Line During Laparoscopic Sleeve Gastrectomy on Early Postoperative Outcomes: A Randomized Trial
Brief Title: Comparison of Omentopexy and Clips on the Staple Line During Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammed Taha Demirpolat, Principal investigator, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Clips - Omentopexy
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Compassion; Bleeding; Nausea, Postoperative; Readmission
Keywords: Bariatric Surgery; clips versus omentopexy; postoperative outcomes
MeSH Terms: conditions — Hemorrhage; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omentopexy with LSG (Active Comparator): We performed omentopexy on staple line after LSG
  Interventions: Procedure: Omentopexy group
- Clips with LSG (Active Comparator): we performed Clips on staple line after LSG
  Interventions: Procedure: Omentopexy group

INTERVENTIONS:
Procedure: Omentopexy group — Omentopexy and Clips on staple line during LSG
  Other Names: Clips group

SUMMARY:
Background: Bleeding through the staple line has been reported as one of the most common staple-related complications in laparoscopic sleeve gastrectomy (LSG). In this study, we aimed to compare the effects of clips and omentopexy techniques on postoperative bleeding and readmissions during the first 30-days following surgery.

Methods: In this prospective randomized controlled study, patients were divided into two groups: clips group and omentopexy group. The groups were compared in terms of postoperative decrease in hemoglobin and hematocrit values, preoperative and peroperative blood pressure values, duration of surgery, number of patients requiring erythrocyte suspension (ES) transfusion, length of hospital stay, hospital readmissions in the first 30-days postoperatively and early postoperative complications.

DETAILED DESCRIPTION:
Study Design and Population This prospective randomized controlled trial was conducted at the University of Health Science Umraniye Training and Research hospital. The Patients who underwent LSG, were between the ages of 18 and 65, with a Body Mass Index (BMI) ≥ 40 or BMI ≥ 35 with at least one obesity-related comorbidity were included in the study. Patients who underwent other bariatric surgery procedures, who declined to be participate in the study, had uncontrolled hypertension, and had preoperative history of gastroesophageal reflux disease (GERD) symptoms were excluded. Approval for the study was received from the ethics committee of tertiary health institution (21.06.2023/218494864). This study is registered on clinicaltrial.gov (). Before the surgery, each of the participants were received comprehensive information about the study, the techniques to be applied were explained, they would be randomly assigned in one of the two groups and the consent form obtained in this context. The CONSORT reporting guidelines were used in this study (17).

Study Groups In the study, patients were divided into two groups: Patients who underwent consecutive clippping along the staple line of the remnant stomach during LSG (clips group) and patients who underwent continuous through-and-through omentopexy of the omentum to the remnant stomach staple line after resection during LSG (omentopexy group).

Data Collection Age, gender, comorbidities, smoking history, preoperative height-weight-BMI values, preoperative systolic blood pressure (SBP)-diastolic blood pressure (DBP) values, preoperative hemoglobin-hematocrit values, peroperative SBP-DBP-mean blood pressure (MBP), duration of surgery, postoperative 6th hour and time of discharge hemoglobin-hematocrit values, number of patients transfused erythrocyte suspension (ES) or requiring invasive intervention due to bleeding, length of hospital stay, hospital readmissions in the first postoperative month, and early postoperative complications were recorded. Duration of surgery was determined from the first skin incision to the last skin suture.

Preoperative, peroperative and Postoperative Evaluation Preoperative anesthesia, cardiology and pulmonology evaluations were performed for each patient. Hepatobiliary ultrasound and upper gastrointestinal endoscopy evaluation were performed. Each patient was administered low molecular weight heparin (enoxaparin 6000 units 1x1 subcutaneously) 12 hours before surgery and was taken to surgery with antiembolism stockings. Intermittant pneumatic compressor device was used perioperatively. Omentopexy was performed with 3-0 V-loc suture (26 mm, V-20 Tapper) and clippping was performed with endo clips II (10 mm, medium/large). Since ERAS protocol was applied in our clinic, no drain was placed in any patient.

At the 4th postoperative hour, all patients were mobilized, intensive respiratory exercise was performed and clear liquid food was started. Complete blood count and C-reactive protein (CRP) laboratory parameters were checked at postoperative 6th, 24th and 48th hour (discharge). Vital parameters were checked every 6 hours postoperatively. Patients who have an acute decrease in hemoglobin value together with a pulse rate of 100 or more per minute and systolic/diastolic blood pressure values below 90/60 mmHg were considered as bleeding and erythrocyte suspension was transfused. Early on the second postoperative day, the patient who could tolerate oral food and did not require additional intervention was discharged.

The primary outcome of the study was to compare the two methods in terms of early postoperative bleeding. The seconder outcome of the study is to compare the groups in terms of duration of surgery, lengh of hospital stay and hospital readmission in the first 30-days postoperatively.

Randomization Patients were numbered according to the order of enrollment and randomly assigned 1:1 to the clips group or the omentopexy group. Allocations were generated using randomly permuted blocks (available at www.randomization.com). All randomization was done by an individual who wasn't included in the study, and the allocations were preserved in sealed envelopes. A research assistant opened the sealed envelope at the beginning of surgery, disclosing the patient's allocation group to the surgeon. The primary surgeon is naturally not blinded to the patient groups and the other surgeon who records and evaluates the data is blinded to the patient groups. All operations were performed laparoscopically by the same surgeon. Considering a 5% alpha margin of error and an 80% confidence interval, power analysis was used to estimate the appropriate sample size for our study, and the results indicated that 68 patients in each group would be adequate.

Comparison of Groups The groups were compared in terms of postoperative decrease in hemoglobin and hematocrit values, preoperative and peroperative blood pressure values, duration of surgery, length of hospital stay, hospital readmissions in the first 30-days postoperatively, early postoperative complications and number of patients requiring ES transfusion.

ELIGIBILITY:
Inclusion Criteria:

* performed Laparoscopic sleeve gastrectomy,
* consent to participate in the study

Exclusion Criteria:

* performed other bariatric procedures,
* uncontrolled hypertension,
* have a gastroesophageal reflux

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Bleeding rates | 3 months
  comparison of groups in terms of bleeding rates in postoperative process

SECONDARY OUTCOMES:
Hospital readmission rates | 3 months
  comparison of groups in terms of postoperative readmission rates in postoperative first month

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Analysis of data and evolution of patients in postoperative process
Supporting Information: SAP, ICF, CSR